CLINICAL TRIAL: NCT07363252
Title: Investigation of REcurrence Mechanisms to Adjuvant osimertINib in Radically Resected EGFR-mutated NSCLC Patients - REMAIN Study
Brief Title: Investigation of REcurrence Mechanisms to Adjuvant osimertINib in Radically Resected EGFR-mutated NSCLC Patients
Acronym: REMAIN
Status: Not yet recruiting | Type: Observational
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Responsible Party: Sponsor
Other Study IDs: GOIRC-03-2024
Record Dates: First submitted 2025-12-10; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: EGFR-mutated NSCLC
Keywords: EGFR-mutated NSCLC; adjuvant osimertinib; Recurrence
MeSH Terms: conditions — Recurrence | interventions — osimertinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Osimertinib — Characterization of the molecular mechanisms of recurrence to adjuvant osimertinib

SUMMARY:
Retrospective-prospective observational multicentric study including radically resected EGFR-mutated NSCLC patients relapsed during or after adjuvant osimertinib, received according to clinical practice

DETAILED DESCRIPTION:
This study will include patients

1. who have already received adjuvant osimertinib and who relapsed at the end of the treatment (off-treatment recurrence) and patients
2. who relapsed during the treatment (on-treatment recurrence). Patients could be enrolled at the time or after the recurrence. Data regarding clinical features for each patient, including demographics and comorbidities, and clinical outcomes of adjuvant osimertinib will be collected.

NGS analysis will be centrally performed on tissue biopsy and/or liquid biopsy collected at the time of recurrence in EGFR-mutated NSCLC treated with adjuvant osimertinib. NGS will be also centrally performed on tissue samples collected at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of radically resected IB-IIIA NSCLC with EGFR activating mutation
* Treatment with adjuvant osimertinib (starting from September 2022, date of approval) according to clinical practice
* Recurrence of disease during or after adjuvant therapy with osimertinib received according to clinical practice
* Availability of tissue and/or liquid biopsy sample collected at the time of recurrence
* Signed informed consent.

  * Exclusion Criteria:
* Unavailability of tissue and/or liquid biopsy sample collected at the time of recurrence
* Concomitant synchronous malignancies aside from NSCLC or any concurrent and/or active malignancy that has required treatment within 2 years
* Involvement in the planning and/or conduct of the study (applies to both investigator staff and/or staff at the study site).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 relapsed EGFR-mutated NSCLC patient receiving osimertinib in adjuvant setting and with tissue biopsy and/or liquid biopsy collected at the time of recurrence
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study is the frequency of new variant(s) detected by Next Generation Sequencing (NGS) Panel at the time of recurrence to adjuvant osimertinib in tissue and/or liquid biopsy | 3 years
  The primary endpoint of the study is the frequency of new variant(s) detected by Next Generation Sequencing (NGS) Panel at the time of recurrence to adjuvant osimertinib in tissue and/or liquid biopsy

SECONDARY OUTCOMES:
Secondary endpoint | 3 years
  • Frequency of new variant(s) in Next Generation Sequencing (NGS) Panel in tissue sample at the time of recurrence to adjuvant osimertinib compared to surgical/pre-osimertinib sample
Secondary endpoint | 3 years
  • percent of treatment options at disease relapse
Secondary endpoint | 3 years
  • Correlation of new variants in NGS and clinical features to the onset of recurrence (on treatment/off treatment)

CONTACTS AND LOCATIONS:
Locations (25):
- Italy (25):
  - IRCCS Oncologico Giovanni Paolo II, Bari, BA
  - Asst Papa Giovanni Xxiii Sc Oncologia, Bergamo, BG
  - UOC di Oncologia Medica IRCCS - Policlinico S. Orsola Malpighi, Bologna, BO
  - Humanitas Istituto Clinico Catanese Contrada Cubba, Misterbianco, CT
  - A.S.S.T - Monza Ospedale San Gerardo, Monza, MB
  - Irccs Humanitas Research Hospital, Milan, MI
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, MI
  - Ospedale San Raffaele Dipartimento di Oncologia Medica, Milan, MI
  - European Institute of Oncology IRCCS, Milan, MI
  - Grande Ospedale Metropolitano Niguarda Ca' Granda, Milan, MI
  - Dip Oncologia-Ematologia - UO Oncologia AOU Policlinico di Modena, Modena, MO
  - UOC di Oncologia Medica 2 - IOV Istituto Oncologico Veneto, Padua, PD
  - S.O.C. di Oncologia Medica e dei Tumori Immuno-correlati, Centro di Riferimento Oncologico IRCCS, Aviano, PN
  - UOC di Oncologia Medica Azienda Ospedaliero-Universitaria di Parma, Parma, PR
  - U.O.C. Oncologia Medica Azienda Unità Sanitaria Locale della Romagna, Ravenna, RA
  - S.C. Oncologia Provinciale, Azienda USL-IRCCS di Reggio Emilia, Reggio Emilia, RE
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma, RM
  - Ifo-Istituto Regina Elena - Oncologia Medica 1, Roma, RM
  - Fondazione Policlinico Universitario 'Agostino Gemelli' IRCCS, Roma, RM
  - AOU San Luigi Gonzaga - SSD oncologia polmonare, Orbassano, TO
  - SC Oncologia ASST Sette Laghi "Ospedale di Circolo e Fondazione Macchi ", Varese, VA
  - "OSPEDALE P. PEDERZOLI" Casa di Cura Privata S.p.A., Peschiera del Garda, VR
  - AOU Integrata di Verona - Ospedale Borgo Trento, Verona, VR
  - Oncologia Clinica Sperimentale Toraco-Polmonare, IRCCS Pascale di Napoli, Napoli
  - A.O.U. "Maggiore della Carita'"- S.C.D.U Oncologia, Novara